CLINICAL TRIAL: NCT04361409
Title: A Phase I Pilot Study of B Cell Depletion With Rituximab Following by Chemotherapy With Cisplatin Plus Gemcitabine for Recurrent Unresectable or Metastatic Head and Neck Cancer Squamous Cell Carcinoma Patients.
Brief Title: Rituximab Plus Chemotherapy in Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Ching Yun Hsieh, attending physician, China Medical University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUH HO-02
Record Dates: First submitted 2013-08-21; First posted 2020-04-24 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Head and Neck Squamous Carcinoma
Keywords: head and neck squamous cell carcinoma; Rituximab; recurrent or metastatic
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Recurrence; Neoplasm Metastasis | interventions — Rituximab; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab plus chemotherapy (Experimental): * Drug:Rituximab
  * Drug:Cisplatin
  * Drug:Gemcitabine
  Interventions: Drug: Rituximab; Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Rituximab — 375mg/m2 on Day-14 and Day-7
  Other Names: Mab thera
Drug: Cisplatin — 70mg/m2 on Day1
  Other Names: Platinex
Drug: Gemcitabine — 1000mg/m2 on Day8
  Other Names: Gemzar

SUMMARY:
Head and neck squamous cell carcinoma (HNSCC) is an important disease with the incidence of 6th all over the world. In Taiwan it is the fifth of male cancer mortality. Most of the patients were middle age and the impact for economy and society was incredible. For recurrent or metastatic HNSCC, the average life span was around 4-6 months. Most patients just can receive chemotherapy. However the chemotherapy can't have any survival benefit. Recently a study showed the Cetuximab plus chemotherapy with cisplatin and 5-fluorouracil had survival benefit in the recurrent or metastatic HNSCC. However in Taiwan, the cetuximab can't be given by health insurance for the patients of the situation.

A lot of investigations recently showed the B lymphocytes got involvements in the squamous cell carcinoma carcinogenesis and tumor progression. In addition the B cell will influence the tumor associated macrophages and myeloid derived suppressor cells. Those immune cells could decrease the affect of chemotherapy and radiotherapy. Thus the B cell depletion has the possibility to develop a new treatment policy. Therefore investigators create a pilot clinical trial using Rituximab plus chemotherapy with cisplatin and gemcitabine for recurrent or metastatic HNSCC.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed squamous cell carcinoma of head and neck.
2. Locoregional recurrence and/or metastases after primary curative local treatment and unsuitable for further radiotherapy and surgery; or primary distant metastases at diagnosis.
3. Measurable disease. Defined as presence of at least one lesion as being ≥10 mm in at least one dimension measured with conventional computed tomography (CT) or ≥10 mm in at least one dimension measured with spiral CT scan or magnetic resonance imaging (MRI)
4. Eastern Cooperative Oncology Group performance status ≤2;
5. Age between 20 and 65 years; and life expectancy of at least 12 weeks.
6. Prior treatments with radiation therapy for palliative management of non-target lesion metastatic disease is permitted provided that at least 2 weeks have relapsed since the last fraction of radiation therapy, disease progression has been documented and all treatment related adverse events are ≦ grade 1 at the time of registration.
7. Negative pregnancy test, Fertile patients must use effective contraception
8. No history of allergic reactions attributed to Rituximab/cisplatin/gemcitabine
9. Patient consent must be obtained

Exclusion Criteria:

1. Presence of central nervous system (CNS) metastases;
2. Presence of other malignancy with the exception of curatively treated non-melanoma skin cancer or cervical carcinoma in situ prior to entry into the study
3. Presence of bone-only metastasis
4. The organ function measured within 14 days prior to study entry as defined below: White blood cell (WBC) less than 2,000/mm3, absolute neutrophil count (ANC) less than 1,500/mm3, or platelets less than 100,000/mm3; serum bilirubin greater than 1.5 times the upper limit of normal range (ULN); alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 2.5 times the ULN if no demonstrable liver metastases, or greater than 5 times the ULN in the presence of liver metastases; creatinine clearance ≤60 ml/min (based upon urine collection);
5. Concomitant illness including uncontrolled infection or other active, uncontrolled disease such as congestive heart failure, angina pectoris, respiratory insufficiency, and arrhythmia.
6. Documented hypersensitivity to platinum compounds or compounds of similar chemical or biologic composition
7. Pregnant or lactating women.
8. Under rituximab treatment or have ever received rituximab within six months.
9. Ongoing other concurrent investigational agents or anticancer therapy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
feasibility of the combination of Rituximab with Gemcitabin/cisplatin in R/M HNSCC | One week after Rituximab and chemotherapy administration.
  Unexpected adverse event. An AE that is not listed in the drug's current labeling, or An AE that is more severe or more specific than indicated in the labeling.

SECONDARY OUTCOMES:
Response rate | through study completion, an average of 1 years
  CT scan according to the RECIST 1.1 criteria.
progression survival | through study completion, an average of 6 months
  The time from the study registration date to the first day of disease progression at any site or of death by any cause.
Adverse event | through study completion, an average of 6 months
  Record adverse event

CONTACTS AND LOCATIONS:
Locations (1):
- China medical University hospital, Taichung, Taiwan

REFERENCES:
- [Derived] Hsieh CY, Lien MY, Lin CY, Lo WJ, Hua CH, Chang WC, Chiu CF, Lin CC. Rituximab in combination with gemcitabine plus cisplatin in patients with recurrent and metastatic head and neck squamous cell carcinoma: a phase I trial. BMC Cancer. 2022 Feb 15;22(1):169. doi: 10.1186/s12885-022-09258-0. PMID 35168547